CLINICAL TRIAL: NCT02850211
Title: A Selective COX-2 Inhibitor Provides Pain Control But Hinders Healing Following Arthroscopic Rotator Cuff Repair: A Prospective Randomized Comparison
Brief Title: A Selective COX-2 Inhibitor Provides Pain Control But Hinders Healing Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Joo Han Oh, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1105/128-003
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Celecoxib; Ibuprofen; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Celecoxib (Experimental): 1 capsule of 200mg Celebrex twice a day for 14 days
  Interventions: Drug: Celecoxib
- Traditional NSAIDs (Active Comparator): 1 tablet of 385mg Ibuprofen twice a day for 14 days
  Interventions: Drug: Ibuprofen
- Opioid drug (Active Comparator): 1 tablet of 50mg Tramadol twice a day for 14 days
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Celecoxib — 1 capsule of 200mg Celebrex PO(per oral) twice a day for 14 days
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Ibuprofen — 1 tablet of 385mg Ibuprofen PO(per oral) twice a day for 14 days
  Other Names: Carol-F
  Arms: Traditional NSAIDs
Drug: Tramadol — 1 tablet of 50mg Tramadol PO(per oral) twice a day for 14 days
  Other Names: Tridol
  Arms: Opioid drug

SUMMARY:
Selective cyclooxygenase (COX)-2 inhibitors are commonly used analgesics that provide similar analgesia but reduced adverse effects compared to other analgesics. However, few studies have been conducted on postoperative pain and tendon-to-bone healing. Here, the investigators investigated the effect of a selective COX-2 inhibitor on analgesia and tendon-to-bone healing following arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Participants Selection After obtaining institutional review board approval and written informed consent from all participants, the investigators prospectively enrolled 180 participants scheduled to undergo arthroscopic acromioplasty and rotator cuff repair for a partial or full thickness tear between September 2011 and August 2012.

A priori statistical power analysis was performed to calculate the number of subjects required. A difference of one point in the visual analogue scale (VAS) was defined as the minimal clinically important difference. With a power of 80% and an alpha of 0.05, the power analysis demonstrated that a sample size of 51 participants per group was needed. Assuming a dropout rate of 20%, the investigators calculated a sample size of 60 participants per group.

Participants were randomly assigned in equal numbers to receive selective COX-2 inhibitors (celecoxib; Celebrex® 200 mg bid, Pfizer, Korea), traditional NSAIDs (ibuprofen; Carol-F® 385 mg tid, Ildong, Korea), or opioid drugs (tramadol; Tridol® 50 mg bid, Yuhan, Korea) for 2 weeks from the first day after surgery.

Analgesic medication was not prescribed preoperatively. Subacromial participant-controlled analgesia (Automed 3200, Ace Medical, Seoul, Korea) was used for the first 48 hours postoperatively in all participants. Intravenous cefazolin was used as the postoperative antibiotic for one day. If participants could not tolerate pain with regular postoperative medication, oxycodone (IR codon 5 mg, Unimed, Korea) was administered as rescue medication; the maximum dosage was limited to 20 mg per day according to the investigators institution's standard postoperative pain control procedures for 2 weeks after surgery.

Clinical and Radiological Assessment Participants rated pain and satisfaction with medication using a VAS of 0 (no pain/no satisfaction) to 10 (unbearable pain/extreme satisfaction) preoperatively and 3 days and 2 weeks postoperatively. Administration of rescue medication and side effects were also recorded. Side effects were categorized into five categories: nausea/vomiting, somnolence/dizziness, gastrointestinal complications (constipation, diarrhea, abdominal discomfort), pruritus, and bruising; respiratory difficulties, renal failure, heart failure, and seizure were also evaluated.

Of the 180 participants, 82 were followed for at least 24 months after surgery. Shoulder functional scores were obtained based on range of motion (ROM) data, pain VAS scores, Constant-Murley Shoulder scores, American Shoulder and Elbow Surgeons scores, and Korean Shoulder Scoring system scores. Radiological integrity of the repaired rotator cuff was assessed using magnetic resonance imaging (MRI) in 70 participants (25 in the celecoxib group, 23 in the ibuprofen group, and 22 in the tramadol group) and ultrasonography in the remaining 12 participants . Postoperative rotator cuff integrity assessed using MRI was categorized as type I to V according to the classification developed by Sugaya et al. as follows: type I, sufficient thickness compared with the normal cuff and homogenously low intensity; type II, sufficient thickness compared with the normal cuff and partial high intensity; type III, insufficient thickness (less than half the thickness of the normal cuff) but no discontinuity, suggesting a partial-thickness delaminated tear; type IV, presence of a minor discontinuity in 1-2 slices on both oblique coronal and sagittal images, suggesting a small full-thickness tear; type V, presence of a major discontinuity in more than two slices on both oblique coronal and sagittal images, suggesting a medium or large full-thickness tear. Postoperative incomplete healing or re-tear was defined as either Sugaya type IV or V.

MRI and ultrasonography data were analyzed by a musculoskeletal radiologist with 10 years of experience who was blinded to the study. The deltoid muscle, subacromial/subdeltoid bursa, long head of the biceps tendon, and entire rotator cuff were examined, with special emphasis on the integrity of the subscapularis tendon, supraspinatus tendon, infraspinatus tendon, and teres minor tendon. The tendons were scanned along their long and short axes. The radiologist defined a full-thickness tear as incomplete healing or a re-tear, such as a hypoechoic full-thickness cleft inside the tendon, detachment of the tendon from the bone, insertion with medial dislocation, and non-visualization of the tendon.

Surgical Procedure and Postoperative Care The senior investigator conducted all surgical procedures arthroscopically using three portals: anterior, lateral, and posterior. In participants with a stiff shoulder, manipulation was performed with capsular release. Synovectomy, biceps procedures, and debridement for partially torn rotator cuff tendons were performed for the glenohumeral joint. After glenohumeral procedures, subacromial decompression was performed to remove inflamed bursal tissue, and acromioplasty was conducted with a motorized burr in almost all participants except those with an extremely thin acromion to yield a flat acromion undersurface and to ensure adequate working space for the repair. Distal clavicle resection was performed in selected participants. The anteroposterior and retraction size of the tear were measured with a calibrated probe, and footprint preparation was performed with a ring curette, rasp, and shaver to expose the bleeding bony surface. After anchors were inserted according to the selected repair technique, the loaded sutures were passed through the tendon using a flexible suture passer (Expressew®, Depuy Mitek, Raynham, MA) or a suture passer (Spectrum®, Linvatec, Largo, FL). All sutures were secured using the SMC knot. After subacromial procedures, the operator always returned to the glenohumeral joint for irrigation and to identify medial anchor pull-out, missed foreign materials, or biceps incorporated into rotator cuff repair.

All participants followed the same rehabilitation protocol. They wore an abduction brace for 5 weeks and started passive ROM after brace removal. Participants who had limited motion preoperatively started tolerable controlled passive motion right after pain had subsided postoperatively. Shrugging of the shoulder and active motion of the elbow (flexion, extension), forearm (supination, pronation), wrist, and hand were encouraged immediately after surgery. After brace weaning, active assisted ROM was performed according to a pre-established protocol for 6 weeks. After full passive ROM was obtained, muscle-strengthening exercises were started; all sports activities were permitted 6 months after surgery. All physical therapy protocols were followed with the cooperation and supervision of a rehabilitation physician.

Statistical Analysis Statistical analysis was performed using SPSS software (version 18.0E; SPSS Inc., Chicago, IL). Frequency and descriptive statistics were analyzed to determine the baseline characteristics, and the t-test, chi-square test, analysis of variance, and Mann-Whitney test were performed to compare the three groups. Tukey's post-hoc test and Bonferroni's test were used to determine the groups between which differences occurred. Statistical significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo arthroscopic acromioplasty and rotator cuff repair for a partial or full thickness tear
* Age < 80 years at time of diagnosis
* Patient willing and able to comply with the study prescriptions
* Patient able to give written informed consent before patient registration/randomisation

Exclusion Criteria:

* Patients with rotator cuff tear arthropathy
* Severe osteoarthritis (Samilson-Prieto grade II or higher)
* Rheumatoid arthritis
* Chronic renal failure (i.e., at high risk for the use of NSAIDs or opioid drugs)
* Liver failure
* Myocardial infarction or chronic heart failure
* Cerebral vascular disease
* Active gastric ulcer or bleeding
* Allergies to NSAIDs or opioid drugs
* Previous surgery on the same side
* Pregnant or breast feeding patients
* Those not willing to participate in the trial

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Rotator cuff healing failure | Day 730
  Assessed by a musculoskeletal radiologist using MRI and ultrasonography

SECONDARY OUTCOMES:
Pain VAS score | Day 0, Day 3, Day 14 Day 730
  Decrease in the VAS (pain in mm) from Day 0 to Day 730
Medication satisfaction VAS score | Day 0, Day 3 and Day 14
  Increase in the VAS (satisfaction in mm) from Day 0 to Day 14
Adverse effects | Day 3 and Day 14
  frequency of adverse effects at Day 3 and Day 14
Constant-Murley Shoulder score | Day 730
American Shoulder and Elbow Surgeons score | Day 730
Korean Shoulder Scoring System | Day 730

CONTACTS AND LOCATIONS:
Overall Officials: Joo Han Oh, MD, PhD, Study Chair — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oh JH, Seo HJ, Lee YH, Choi HY, Joung HY, Kim SH. Do Selective COX-2 Inhibitors Affect Pain Control and Healing After Arthroscopic Rotator Cuff Repair? A Preliminary Study. Am J Sports Med. 2018 Mar;46(3):679-686. doi: 10.1177/0363546517744219. Epub 2017 Dec 18. PMID 29253346